CLINICAL TRIAL: NCT05890040
Title: Evaluation of the Effect of Watching Surgery Videos on Social Media on Anxiety Before Impacted Wisdom Tooth Extraction
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Berkan Altay, DDS, Principal Investigator, Kutahya Health Sciences University
Other Study IDs: 021/12-08
Record Dates: First submitted 2023-03-28; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Impacted Wisdom Teeth
Keywords: Social media; surgery video
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients watching surgery video: Situational and trait anxiety test will be applied to patients.
  Interventions: Other: questionnaire
- patients who did not watch the surgery video: Situational and trait anxiety test will be applied to patients.
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — assessment of anxiety

SUMMARY:
Surgical extraction of impacted wisdom teeth creates a high level of anxiety on patients. Anxiety in patients can affect the difficulty of tooth extraction, prolong the duration of surgery and increase post-operative pain. With the increasing internet usage in recent years; patients can access different information about surgical procedures by watching videos on various social media platforms in an uncontrolled manner. In the literature, the effects of impacted tooth extraction videos, which are watched by physicians before the operation, on anxiety have been examined. However, studies on the evaluation of the effect of the surgery videos watched by the patients before the surgery on their own will on anxiety and pain perception have been limited.

DETAILED DESCRIPTION:
The study is given to KSBU Faculty of Dentistry, Department of Oral, Dental and Maxillofacial Surgery; It will be applied to patients who are referred from Oral, Dental and Maxillofacial Radiology and who want to participate in the study. In our study, the Situational-Trait Anxiety Inventory will be used to assess anxiety. Patients who are referred to our clinic from Oral, Dental and Maxillofacial Radiology and who have impacted wisdom teeth will be evaluated in terms of extraction indication. Patients with indications for extraction will be asked to rate the sentences in the State and Trait Anxiety Inventory when making an appointment. Patients will be informed about impacted tooth extraction as it is routinely practiced. Within the scope of this study, no information about the extraction will be given in the Oral, Dental and Maxillofacial Radiology clinic, standard information will be given to the patients in our clinic and the surgery appointment will be given one week later. On the day of tooth extraction, patients will be asked whether they watched a video about impacted tooth extraction from any social media platform. The patients who watch the video will be assigned to the study group, and the patients who do not watch the video will be assigned to the control group, so the study will be conducted over two groups. If the patient has watched the video; He will be asked whether he watches an animation video or a video with real surgery footage, and the reason for watching the video. Then, before starting the operation, they will be asked to score the sentences in the Situational and Trait Anxiety Inventory. By comparing the Situational Anxiety Inventory made at the time of the surgery appointment with the Situational Anxiety Inventory scores made just before the surgery, it will be evaluated whether the patients who watch videos have more anxiety. At the same time, it will be evaluated whether the patients who have a high Trait Anxiety Inventory score when making an appointment and who generally have high anxiety watch more videos. This study is planned to be performed on a total of 60 patients, 30 of whom watch videos and 30 who do not.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-45
* The patient does not have any systemic disease.
* Patients with mesio-angular or 2 or 3 / B according to the Pell and Gregory classification of the impacted tooth radiographic grade according to Winter classification

Exclusion Criteria:

* Patients using antidepressant and anxiolytic drugs
* Patients with a history of impacted tooth extraction/difficult tooth extraction
* Patients with systemic disease
* Female patients who are pregnant or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients between the ages of 18-45 who want to have their impacted tooth extracted
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2023-07-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of anxiety in impacted wisdom tooth extraction | one week before impacted tooth extraction
  State and trait anxiety inventory( STAI-T and STAI-S)
Evaluation of anxiety in impacted wisdom tooth extraction | just before impacted tooth extraction
  State and trait anxiety inventory( STAI-T and STAI-S)

CONTACTS AND LOCATIONS:
Overall Officials: Berkan Altay, DDS, Principal Investigator — 05356557441
Locations (1):
- Kutahya University of Health Sciences, Kütahya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/40/NCT05890040/Prot_SAP_ICF_000.pdf